CLINICAL TRIAL: NCT03826472
Title: Almond Butter and Fasting Glucose in Adults With Type 2 Diabetes
Brief Title: Almond Butter and Fasting Glucose
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PKE AlmondButter
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Almond Butter (Experimental): Participants will consume one ounce per day (~32 g) of almond butter as an evening snack (i.e., after dinner and before sleep).
  Interventions: Other: Almond Butter
- No-snack Control (No Intervention): Participants will consume nothing besides water after dinner/bed sleep.

INTERVENTIONS:
Other: Almond Butter — Natural almond butter
  Arms: Almond Butter

SUMMARY:
A two-period randomized crossover study will be conducted to determine the effect of almond butter as an evening snack on fasting blood glucose in adults with type 2 diabetes, not taking insulin.

DETAILED DESCRIPTION:
Control of fasting blood glucose is a challenge for many individuals with diabetes. Researchers want to better understand how a nighttime snack can affect morning fasting blood glucose. A two-period randomized crossover trial will be conducted. Participants will be randomized to receive each treatment for 1 week. During the almond butter treatment, participants will consume 2 tbsp of almond butter per day as an evening snack. The control treatments will be a no-snack control. Fasting blood glucose, as well as glucose trends, will be measured using Continuous Glucose Monitor (CGM). Participants will also be asked to take simple cognitive tests on a study-provided smartphone each day of the study and report their daily food intake and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with diagnosed type 2 diabetes
* Not on insulin therapy
* On stable does of oral antihyperglycemic agent (no dose change for 6 months)
* Currently monitoring blood glucose at home via glucometer
* Willing and able to adhere to study protocol

Exclusion Criteria:

* Individuals with type 1 diabetes, cardiovascular disease, kidney disease, liver disease, cancer or inflammatory conditions (e.g. GI disorders, rheumatoid arthritis)
* Women who are pregnant, breastfeeding, or have been pregnant within the last 6 months or breastfeeding within the last 6 weeks
* Individuals who smoke or use tobacco products
* Use of insulin therapy or sulfonylurea medications
* Allergy to any tree nut
* Liver or kidney disease
* Allergy to Dexcom CGM adhesive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, RDN, Principal Investigator — Penn State
Locations (1):
- Penn State, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a crossover study, a total of 10 participants completed the study. Data from 1 participant was not used due a technology issue.
Groups:
- Almond Butter-No Snack Control: First intervention:
  Participants will consume one ounce per day (~32 g) of almond butter as an evening snack (i.e., after dinner and before sleep).
  Almond Butter: Natural almond butter
  Second intervention:
  Participants will consume nothing besides water after dinner/bed sleep.
- No-snack Control-Almond Butter: First intervention:
  Participants will consume nothing besides water after dinner/bed sleep.
  Second intervention:
  Participants will consume one ounce per day (~32 g) of almond butter as an evening snack (i.e., after dinner and before sleep).
  Almond Butter: Natural almond butter
Period: First Intervention (1-week)
Arm/Group | Almond Butter-No Snack Control | No-snack Control-Almond Butter
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention (1-week)
Arm/Group | Almond Butter-No Snack Control | No-snack Control-Almond Butter
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Almond Butter-No Snack: First intervention:
  Participants will consume one ounce per day (~32 g) of almond butter as an evening snack (i.e., after dinner and before sleep).
  Almond Butter: Natural almond butter
  Second intervention:
  Participants will consume nothing besides water after dinner/bed sleep.
- No Snack-Almond Butter: First intervention:
  Participants will consume nothing besides water after dinner/bed sleep.
  Second intervention:
  Participants will consume one ounce per day (~32 g) of almond butter as an evening snack (i.e., after dinner and before sleep).
  Almond Butter: Natural almond butter
- Total: Total of all reporting groups
Arm/Group | Almond Butter-No Snack | No Snack-Almond Butter | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Full Range); unit: years] | 59 [53 to 73] | 58 [42 to 71] | 58 [42 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10
Mean duration of diabetes [Mean (Full Range); unit: years] | 8.2 [3 to 15] | 6.8 [1 to 14] | 7.5 [1 to 15]
Home self-monitoring of blood glucose prior to study start [Count of Participants; unit: Participants] | 1 | 5 | 6
Medication use [Number; unit: participants] | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Fasting Glucose Measured Using Continuous Glucose Monitoring
Description: Fasting glucose measures how much glucose (sugar) is in a blood sample after an overnight fast. In this study, fasting glucose was measured by continuous glucose monitoring (interstitial glucose); fasting window identified through review of glucose monitoring data to be 4am-6am.
Time Frame: 2 weeks
Population: Adults with a diagnosis of type 2 diabetes, not on insulin therapy.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Almond Butter: Participants instructed to consume study provided 2 tbsp of natural almond butter after dinner and before bed.
- No-snack Control: Participants asked not to consume any food or beverages besides water after dinner.
Arm/Group | Almond Butter | No-snack Control
Number analyzed (Participants) | 9 | 9
mg/dL | 148.6 [94.9 to 202.3] | 142.1 [94 to 190.3]

2. Secondary Outcome: Glucose Trends
Description: Overnight (12pm-4am) mean blood sugar values measured by continuous glucose monitoring (interstitial glucose)
Time Frame: 2 weeks
Population: 9 participants total; 9 analyzed in each group (crossover study)
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Almond Butter | No-snack Control
Number analyzed (Participants) | 9 | 9
mg/dL | 147.7 [92.6 to 202.8] | 142.2 [91.8 to 191]

3. Secondary Outcome: Inhibitory Control Task (Percent Correct)
Description: Go-NoGo task asked participants to press a button when a letter other than X was on screen and not press a button when X was present.
Time Frame: 2 weeks
Population: 9 participants total; 9 analyzed in each group (crossover study)
Measure: Mean (Standard Deviation); unit: percentage correct
Groups:
- Almond Butter: Participants instructed to consume study provided 2 tbsp of natural almond butter
- No Snack Control: Participants asked not to consume any food or beverages besides water after dinner.
Arm/Group | Almond Butter | No Snack Control
Number analyzed (Participants) | 9 | 9
percentage correct | 35.34 (1.51) | 35.51 (1.98)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Groups:
- Almond Butter: 2 tbsp of natural almond butter measured out and provided by metabolic kitchen to be consumed after dinner and before bed
- No-snack Control: Participants asked not to consume any food or beverage besides water after dinner (unless medically necessary)
Arm/Group | Almond Butter | No-snack Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was a pilot study; interpretation of results is limited by small sample size and short study duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT03826472/Prot_SAP_002.pdf